CLINICAL TRIAL: NCT03313752
Title: Study on the Effect of Dapagliflozin on Myocardial Insulin Sensitivity and Perfusion
Brief Title: Effects of SGLT2 Inhibition on Myocardial Insulin Sensitivity
Acronym: DapaHeart
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andrea Giaccari (Other)
Responsible Party: Sponsor-Investigator, Andrea Giaccari, Associate Professor, Catholic University of the Sacred Heart
Organization: Catholic University of the Sacred Heart (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-003614-27
Record Dates: First submitted 2017-10-04; First posted 2017-10-18 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Type2 Diabetes Mellitus; Stable Coronary Artery Disease
Keywords: diabetes, heart, dapagliflozin,
MeSH Terms: conditions — Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A - placebo (Placebo Comparator): Green, plain, diamond shaped, film coated tablet (orally), not containing active ingredient; once daily, for 4 weeks
  Interventions: Other: Placebo
- B - experimental drug (Experimental): Dapagliflozin tablet available at dose of 10 mg, once daily, for 4 weeks
  Interventions: Drug: Dapagliflozin 10Mg Tab

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — Dapagliflozin, will be administered according to the approved posology and to the approved dose as stated by Local Health Indication and by the Drug Brochure
  Arms: B - experimental drug
Other: Placebo — placebo
  Arms: A - placebo

SUMMARY:
A Phase III, single-centre, randomized, 2-arm, parallel-group, double blind, placebo-controlled study, consisting of a screening phase (Days -14 to -1), a 4-week double-blind, placebo-controlled treatment phase and a 4-week follow-up phase.

Subjects: Type 2 diabetic patients and coronary artery diseases (CAD) not requiring revascularization or underwent percutaneous coronary intervention (PCI) but clinically stable at time of screening visit, with suboptimal glycaemic control (HbA1c 7.0-8.5%) on their current anti-hyperglycaemic regimen

Subjects will be randomized in a 1:1 ratio to dapagliflozin or placebo.

Subjects will undergo screening assessment in the 14-day period preceding administration of the first dose of study drug on Day 1.

The primary Objective is to assess the effect of dapagliflozin on myocardial insulin sensitivity The Secondary Objective is to assess global heart function, and metabolic systemic effects of dapagliflozin, and glycemic control.

The study aims to enroll patients with type 2 diabetes with suboptimal glycemic control, and with coronary artery diseases (CAD) not requiring revascularization or underwent percutaneous coronary intervention (PCI) but clinically stable, who have already undergone, under routine cardiological assessment, a positron emission tomography (PET) 13NH3 scan in order to assess the cardiovascular function. Thus, the study aims to assess whether the improvement in cardiac metabolism obtained with dapagliflozin is greater than that obtained with normal clinical practice (according to Standards of Care).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study-specific procedures
2. Female or male subjects aged between 40 and 75 inclusive. Patients who have been surgically sterilized (hysterectomy or tubal-ligation) at least 12 months prior to screening, or are postmenopausal having had no regular menstrual bleeding for at least one (1) year prior to screening. Menopause will be confirmed by a plasma follicle stimulating hormone (FSH) level of > 35 IU/mL at screening, or Women with childbearing potential willing not to initiate pregnancy during the course of the study, and non-nursing women.

   Men having relationships with women with childbearing potential willing not to procure a pregnancy during the course of the study;
3. Patients with type 2 diabetes
4. Patients with established, stable CAD, defined as ≥30% coronary stenosis in at least one major coronary vessel on invasive coronary angiography (ICA) or computed tomography angiography (CTA) performed within 12 months from screening and no indication to revascularization or with no evidence of critical restenosis, if previously subjected to percutaneous coronary intervention (PCI) (>6months).
5. Patients with a clinical indication for 13N-ammonia PET-CT, as established by a cardiologist, nuclear medicine physician or diabetologist.
6. Patients with a body mass index (BMI) equal or greater than 25 kg/m2 but less than 35 kg/m2 [BMI = Weight (kg) / Height squared (m2)]
7. Patients with a HbA1c between 7.0% and 8.5%, according to the actual clinical conditions of the patients;
8. Patients with diabetes duration <10 years;
9. Patients with stable medical therapy [including other anti-hyperglycemic agents (see Table 1, section 5.2.1 for all therapies allowed, as per current standard treatment); pioglitazone and basal-bolus insulin treatment are excluded, as reported in the exclusion criteria 15] for at least 3 months prior to the screening visit (including stable insulin dose defined as no variation more than 30% in daily insulin dose within the preceding 3 months.
10. Patients with Fasting C-peptide > 1 ng/mL (0.33 nmol/L) at Visit 0

Exclusion Criteria:

1. Type 1 diabetes (as assessed by medical history); previous diagnosis of Latent Autoimmune Diabetes of Adults (LADA), and or not fulfilling inclusion criteria #10
2. History of diabetic ketoacidosis or hyperosmolar non-ketotic coma
3. NYHA class III or IV
4. Unstable angina
5. Previous re-vascularisation (either percutaneous coronary intervention or coronary artery bypass graft) in the last <6 months before screening
6. Reduced left ventricular ejection fraction (≤ 50%)
7. Increased likelihood of developing diabetic ketoacidosis (history of DKA, alcohol consumption, volume depletion dehydration, clinical conditions causing diarrhea, vomit and anorexia)
8. Moderate to severe renal impairment (eGFR<60 ml/min/1.73m2 as calculated by the modification of diet in renal disease [MDRD] equation or end-stage renal disease); overt proteinuria, defined as Spot urine Microalbumin/Cr ratio of >300 mg/g at screening (Visit 0)
9. Severe liver dysfunction
10. Asthma
11. Uncontrolled blood pressure
12. Symptomatic tachy- or bradyarrhythmias
13. Previous acute myocardial infarction
14. Contraindications to adenosine: known hypersensitivity to adenosine or to any of the excipients; sick sinus syndrome, second or third degree atrio-ventricular block (except in patients with a functioning artificial pacemaker); chronic obstructive lung disease with evidence of bronchospasm (e.g. bronchial asthma ); long QT syndrome; severe hypotension; decompensated states of heart failure
15. Use of pioglitazone; use of loop diuretics; basal-bolus insulin therapy; use of systemic steroids less than 3 days prior to the screening visit (Visit 0)
16. Known hypersensitivity to the active substance or to any of the excipients in study drug
17. Inability to provide informed consent
18. Participation in another clinical study with an investigational product during the previous 30 days
19. Patients with history of breast, bladder and prostate cancer
20. Patients who will undergo surgical procedures
21. Patients with acute urinary tract infection
22. Patients with history of intolerance to galactose and lactose
23. Severe/uncontrolled medical conditions, causing liquid volume depletion

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Effect of dapagliflozin on myocardial insulin sensitivity | 4 weeks
  Myocardial Glucose Uptake (MGU) umol/min/gr during euglycemic hyperinsulinemic clamp: change from baseline

SECONDARY OUTCOMES:
Effect on Coronary flow reserve [Main Secondary Outcome] | 4 weeks
  Coronary flow reserve (CFR) obtained as ratio of myocardial blood flow (ml/min/g) (MBF) during pharmacological stress and MBF at rest: change from baseline
3. Browning of white adipose tissue: change from baseline | 4 weeks
  Quantitative measurement of FDG uptake in pericardial, perirenal, interscapular fat by total body FDG PET-CT study, expressed as maximum Standard Uptake Volume (SUVmax) (change from baseline)
Metabolic systemic effects of dapagliflozin | 4 weeks
  Whole body glucose uptake calculated as mg/kg/min during the euglycemic hyperinsulinemic clamp: change from baseline
Effect on Left Ventricular Ejection Fraction at rest | 4 weeks
  Whole body glucose uptake calculated as mg/kg/min during the euglycemic hyperinsulinemic clamp: change from baseline
Effect on Left Ventricular Ejection Fraction during pharmacological stress | 4 weeks
  Left Ventricular Ejection Fraction (percent %) measured by Gated-PET with 13N-ammonia during pharmacological stress: change from baseline
Fasting glucose concentration change from baseline | 4 weeks
  Measured as fasting glucose concentration (mg/dl): change from baseline
Glycemic control change from baseline | 4 weeks
  Measured as Glycated hemoglobin (HbA1c) (percent %): change from baseline
Gut microbiota composition change from baseline | 4 weeks
  Analysis of gut microbiota composition at class, genus, and species levels: change from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Center For Endocrine and Metabolic Diseases - Catholic University, Rome, RM, Italy

REFERENCES:
- [Derived] Cinti F, Leccisotti L, Sorice GP, Capece U, D'Amario D, Lorusso M, Gugliandolo S, Morciano C, Guarneri A, Guzzardi MA, Mezza T, Capotosti A, Indovina L, Ferraro PM, Iozzo P, Crea F, Giordano A, Giaccari A. Dapagliflozin treatment is associated with a reduction of epicardial adipose tissue thickness and epicardial glucose uptake in human type 2 diabetes. Cardiovasc Diabetol. 2023 Dec 19;22(1):349. doi: 10.1186/s12933-023-02091-0. PMID 38115004
- [Derived] Capece U, Pavanello C, Cinti F, Leccisotti L, Mezza T, Ciccarelli G, Moffa S, Di Giuseppe G, Soldovieri L, Brunetti M, Giordano A, Giaccari A, Calabresi L, Ossoli A. Dapagliflozin-Induced Myocardial Flow Reserve Improvement is not Associated with HDL Ability to Stimulate Endothelial Nitric Oxide Production. Diabetes Ther. 2024 Jan;15(1):257-268. doi: 10.1007/s13300-023-01491-5. Epub 2023 Oct 26. PMID 37883003
- [Derived] Leccisotti L, Cinti F, Sorice GP, D'Amario D, Lorusso M, Guzzardi MA, Mezza T, Gugliandolo S, Cocchi C, Capece U, Indovina L, Ferraro PM, Iozzo P, Crea F, Giordano A, Giaccari A. Dapagliflozin improves myocardial flow reserve in patients with type 2 diabetes: the DAPAHEART Trial: a preliminary report. Cardiovasc Diabetol. 2022 Sep 3;21(1):173. doi: 10.1186/s12933-022-01607-4. PMID 36057768
- [Derived] Sorice GP, Cinti F, Leccisotti L, D'Amario D, Lorusso M, Guzzardi MA, Mezza T, Cocchi C, Capece U, Ferraro PM, Crea F, Giordano A, Iozzo P, Giaccari A. Effect of Dapagliflozin on Myocardial Insulin Sensitivity and Perfusion: Rationale and Design of The DAPAHEART Trial. Diabetes Ther. 2021 Jul;12(7):2101-2113. doi: 10.1007/s13300-021-01083-1. Epub 2021 May 26. PMID 34037951